CLINICAL TRIAL: NCT03602040
Title: A Psychoeducational Intervention Supporting Patients With a New Diagnosis and/or Genetic Carrier Status for an Inherited Cardiac Condition-a Feasibility Study
Brief Title: A Psychoeducational Intervention Supporting Patients With an Inherited Cardiac Condition
Acronym: PISICC
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting advice from R&D regarding recruitment
Sponsor: King's College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); King's College Hospital NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 249303; ICA-CDRF-2015-01-046 (Other Grant/Funding Number: National Institute for Health Research); GFWKBQR (Other Grant/Funding Number: Sponsor Number)
Record Dates: First submitted 2018-06-26; First posted 2018-07-26 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Inherited Cardiac Conduction Disorder; Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: This feasibility study will be using mixed methods and will be conducted in 2 phases.Phase 1 of the study is an uncontrolled clinical trial of the psychoeducational education. Phase 2 is a nested qualitative component of the feasibility study and will be comprise of at least 7 semi-structured interviews lasting up to 30 minutes with patients who participated in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PISICC group (Experimental): Psychoeducational intervention
  Interventions: Behavioral: PISICC

INTERVENTIONS:
Behavioral: PISICC — PISICC consists of:
  1. Standard disease-specific information leaflet
  2. Personalised lifestyle consideration form
  3. 1-hour group session with up to 10 participants facilitated by the PhD student who is also an experienced cardiac genetic nurse. This will include discussions of 2 scenarios (communicating with clinicians and communicating with family) and a question and answer session based on the personalised lifestyle consideration form Components a) and b) will be given to the patient after the baseline assessment and there will be an interval of 2 weeks before the participants attend for component c).

SUMMARY:
Inherited heart conditions (IHCs) can cause young sudden deaths due to a genetic trait that leads to a thickened heart muscle or abnormal heart rhythms. Relatives of an affected person have a 50% chance of inheriting IHCs and this is determined either through a blood test (predictive genetic test) and/or physical tests such as a heart tracing (electrocardiogram), scan (echocardiogram) and exercise test. When patients find out they are affected or are carriers for an IHC, they have numerous questions about medical management, prognosis, lifestyle; as well as experiencing stress and anxiety because of the impact on their health and risk to their family. Based on published studies and interviews, a psychoeducational intervention underpinned by Self-determination Theory was developed to support these patients An uncontrolled study to determine the feasibility of the intervention and outcome measures will be undertaken. Patients with a new IHC diagnosis or a carrier result aged 16 years and older will be recruited from outpatient clinics in London and will be receive the intervention consisting of a disease-specific information leaflet, a personalised lifestyle consideration guide and participation in a 1-hour group session facilitated by a cardiac genetic nurse. Outcome measures to look at degree of self-determination, autonomy support and competence; and heart-related anxiety will be collected at baseline and at 3 months post intervention. Clinical and socio-demographic data will be obtained from medical notes. The feasibility and acceptability of the intervention will be measured by assessment of the study procedures such as recruitment, retention and any adverse events. It is expected that there will be up to 4 consecutive group sessions and feedback from each session will be used to co-design and refine the intervention model for a definitive clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are aged 16 and older.
2. Patients who have undergone cardiac screening and/or predictive genetic testing for inherited cardiac conditions and are within 6 months of receiving a new diagnosis of an inherited cardiac condition (ICC) and/or have been found to be carriers of a genetic alteration that can cause an ICC.

Exclusion Criteria:

1. Patients who were initially referred to the clinic for reasons other than cardiac screening and/or predictive genetic testing for ICCs.
2. Patients who have undergone cardiac screening and/or predictive genetic testing for ICCs and more than 6 months have passed since receiving a new diagnosis of an ICC and/or a carrier result for a genetic alteration that can cause an ICC.
3. Patients who have undergone cardiac screening and/or predictive genetic testing for ICCs and have received a negative result.
4. Patients below 16 years of age.
5. Patients with insufficient command of written and spoken English to comprehend study documents and participate in the study procedures and discussion.
6. Patients who are already participating in a study involving a psychoeducational intervention, novel cardiac medication or device.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Engagement of clinical staff with identification of patients | 3 months
  Number of participants identified for recruitment
Engagement of participants with recruitment procedures | 3 months
  Number of participants consented, number of participants declined and withdrawn
Completion of data collection | 3 months
  Rates of data collection at baseline and follow-up, and reasons for missing data
Engagement with psychoeducational intervention | 3 months
  Rates of intervention uptake and reasons for dropout

SECONDARY OUTCOMES:
Perceived Competence Scale | Measured at baseline and 3 months post intervention
  A short 4-item questionnaire assessing feelings of competence about a specific domain. In this case, this is for the management of the diagnosis or carrier status. The score ranges from 28 (high perceived competence) to 4 (low perceived competence) Metric for summarising data: t-test
Perceived Choice and Awareness of Self Scale | Measured at baseline and 3 months post intervention
  A short, 10-item scale, with two 5-item subscales pertaining to perception of choice in one's actions and awareness of oneself. The total score ranges from 50 (high perceived choice and awareness of self) to 10 (low perceived choice and awareness of self). For the perceived choice subscale, the score ranges from 25 (high perceived choice) to 5 (low perceived choice). For the perceived awareness of self subscale, the score ranges from 5 (high perceived awareness of self) to 1 (low perceived awareness of self) Metric for summarising data: t-test
Health Care Climate Questionnaire | Measured at baseline and 3 months post intervention
  A 15-item questionnaire to assess the patients' perception of the degree to which their health care team is supporting their autonomy. The average score ranges from 7 (high perceived autonomy support from clinicians) to 1 (low perceived autonomy support from clinicians).
  Metric for summarising data: t-test
Heart-related Anxiety (Questionnaire) | Measured at baseline and 3 months post intervention
  Cardiac Anxiety Questionnaire-an 18-tem self-reported questionnaire designed to measure heart-focused anxiety. The total score ranges from 72 (high heart-related anxiety) to 0 (low heart-related anxiety) Metric for summarising data: t-test

OTHER OUTCOMES:
Process evaluation (Qualitative interviews) | 3 months
  Nested qualitative component of the study consisting of semi-structured interviews with a subset of patients who participated in the study. The topic guide will gather insights on the patient experience of the intervention and trial procedures. All interviews will be digitally recorded, transcribed and thematic analysis will be facilitated by NVivo software.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Patch, PhD, Principal Investigator — King's College London
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided